CLINICAL TRIAL: NCT04648137
Title: Circulating Oxytocin Changes in Response to the Oxytocin System Stimulator MDMA in Patients With Diabetes Insipidus and Healthy Controls
Acronym: OxyMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2020-02147; me20ChristCrain4
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Insipidus
Keywords: central diabetes insipidus; oxytocin levels; 3,4-methylenedioxymethamphetamine (MDMA); hypothalamic-pituitary axis; hypopituitarism; vasopressin
MeSH Terms: conditions — Diabetes Insipidus; Diabetes Insipidus, Neurogenic; Hypopituitarism

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, cross-over (MDMA versus placebo, within subject comparison) study in patients with central diabetes insipidus versus healthy controls (between-subject comparison). Participants will be randomized to receive either first placebo or first MDMA, respectively.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with central diabetes insipidus (Experimental)
  Interventions: Diagnostic Test: study intervention: 3,4-methylenedioxymethamphetamine (MDMA, ecstasy); Diagnostic Test: Control intervention: Placebo
- Healthy volunteers (Experimental)
  Interventions: Diagnostic Test: study intervention: 3,4-methylenedioxymethamphetamine (MDMA, ecstasy); Diagnostic Test: Control intervention: Placebo

INTERVENTIONS:
Diagnostic Test: study intervention: 3,4-methylenedioxymethamphetamine (MDMA, ecstasy) — single administration of MDMA (100mg): 3,4-methylenedioxymethamphetamine (MDMA, ecstasy) will be prepared as gelatin capsules with mannitol as the filler. MDMA will be administered in a single absolute dose of 100 mg corresponding to a medium high dose of (mean ± SD) 1.3 ± 0.3 mg/kg body weight.
Diagnostic Test: Control intervention: Placebo — Identical placebo (only mannitol) capsules

SUMMARY:
This study is to evaluate oxytocin levels in response to MDMA administration as compared to placebo in patients with diabetes insipidus and healthy volunteers.

DETAILED DESCRIPTION:
Disruption of the hypothalamic-pituitary axis due to congenital abnormalities, tumors or head trauma may cause anterior and/or posterior pituitary deficiency also known as partial or panhypopituitarism. Patients with hypopituitarism, especially those with panhypopituitarism (i.e., anterior and posterior insufficiency) often report residual symptoms and lower quality of life despite adequate substitution treatment of deficient pituitary hormones. A recent study identified a potential oxytocin deficient state in men with combined anterior and posterior deficiency. Due to the close proximity of vasopressin and oxytocin, disruption of the vasopressin system leading to diabetes insipidus could as well disturb the oxytocin system leading to low oxytocin levels. It is therefore possible that the increased psychopathology and reduced quality of life as observed in patients with central diabetes insipidus is caused by an oxytocin deficiency. Several studies documented marked acute increases in circulating oxytocin levels in response to 3,4-methylenedioxymethamphetamine (MDMA) administration as compared to placebo in healthy volunteers.

MDMA could therefore be useful as a provocation test to detect an oxytocin deficiency in patients with central diabetes insipidus. This study is to investigate if oxytocin provocation following a single dose administration of MDMA is reduced in patients with central diabetes insipidus as compared to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria diabetes insipidus:

* Confirmed diagnosis of central diabetes insipidus

Inclusion criteria healthy volunteers:

* Matched for age, sex, BMI and estrogen replacement/menopause/hormonal contraceptives to patients with central diabetes insipidus
* No medication, except hormonal contraception-

Exclusion Criteria:

* Familial central diabetes insipidus
* Participation in a trial with investigational drugs within 30 days
* Illicit substance use (with the exception of cannabis) more than 10 times in lifetime or any time within the previous two months
* Consumption of alcoholic beverages >15 drinks/week
* Tobacco smoking >10 cigarettes/day
* Cardiovascular disease (coronary artery disease, heart failure, left ventricular ejection fraction ( LVEF) <40%, stroke in the last 3 months, atrial fibrillation/flatter, Wolff-Parkinson-White syndrome (WPW)-Syndrome)
* Uncontrolled arterial hypertension (>140/90 mmHg) or hypotension (syst blood pressure <85mmHg)
* Current or previous major psychiatric disorder (e.g., major depression, schizophrenia spectrum disorder)
* Psychotic disorder in first-degree relatives
* Regular intake of selective serotonin reuptake inhibitor (SSRI), monoamine oxidase (MAO)-Inhibitors
* Pregnancy and breastfeeding
* Diagnosed chronic kidney disease (CKD) > grade III (GRF < 30ml/min)
* Diagnosed liver cirrhosis or alanine aminotransferase (ALAT) or aspartate aminotransferase (ASAT) levels 2.5 times above the normal range

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
area under the concentration time curve in oxytocin level | from baseline oxytocin measurement (before intake) to 6 hours after administration of MDMA
  area under the concentration time curve in oxytocin level from baseline oxytocin measurement (before intake) to 6 hours after a single administration of MDMA (100mg) as compared to placebo in the same subjects between patients with central diabetes insipidus and healthy volunteers.

SECONDARY OUTCOMES:
Peak change in oxytocin (OT) plasma level | from baseline oxytocin measurement (before intake) to 6 hours after administration of MDMA
  Peak change in OT plasma level
Time course of plasma OT levels | from baseline oxytocin measurement (before intake) to 6 hours after administration of MDMA
  Time course of plasma OT levels
Time course of plasma MDMA concentration | from baseline oxytocin measurement (before intake) to 6 hours after administration of MDMA
  Time course of plasma MDMA concentration
Time course of cortisol levels | from baseline oxytocin measurement (before intake) to 6 hours after administration of MDMA
  Time course of cortisol levels
Time course of prolactin levels | from baseline oxytocin measurement (before intake) to 6 hours after administration of MDMA
  Time course of prolactin levels
Time course of copeptin levels | from baseline oxytocin measurement (before intake) to 6 hours after administration of MDMA
  Time course of copeptin levels
Time course of adrenocorticotropic hormone (ACTH) levels | from baseline oxytocin measurement (before intake) to 6 hours after administration of MDMA
  Time course of ACTH levels
Subjective/emotional effects | from baseline oxytocin measurement (before intake) to 6 hours after administration of MDMA
  Subjective/emotional effects assessed on a 10-point visual analog scale (e.g., feelings of anxiety, pleasure, fear, 0 = better outcome,10 = worst outcome)
Recognition of negative emotions in the face emotion recognition task (FERT) | from baseline oxytocin measurement (before intake) to 6 hours after administration of MDMA
  Recognition of negative emotions in the face emotion recognition task (FERT)
Empathy in the multifaceted empathy task (MET) | from baseline oxytocin measurement (before intake) to 6 hours after administration of MDMA
  Empathy in the multifaceted empathy task (MET)
Anxiety level with the State-Trait Anxiety Inventory (STAI) | from baseline oxytocin measurement (before intake) to 6 hours after administration of MDMA
  Anxiety level with the State-Trait Anxiety Inventory (STAI)
Level of Alexithymia using the Toronto-Alexithymia-Scale 20 (TAS-20) | from baseline oxytocin measurement (before intake) to 6 hours after administration of MDMA
  Level of Alexithymia using the Toronto-Alexithymia-Scale 20 (TAS-20); total scores can range from 20-100, with higher scores indicating greater impairment/challenges
Level of depression using the Beck-Depressions-Inventory II (BDI-II) | from baseline oxytocin measurement (before intake) to 6 hours after administration of MDMA
  Level of depression using the Beck-Depressions-Inventory II (BDI-II); 21-question multiple-choice self-report inventory. Higher total scores indicate more severe depressive symptoms.
Level of general physical & mental health using the short form health survey (SF-36) | from baseline oxytocin measurement (before intake) to 6 hours after administration of MDMA
  Level of general physical & mental health using the short form health survey (SF-36); 36-item, patient-reported survey of patient health; the higher the score, the more favourable the health state.

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. Dr. med., Principal Investigator — Endocrinology, Diabetes and Metabolism, University Hospital Basel
Locations (1):
- University Hospital Basel, Endocrinology, Diabetes and Metabolism, Basel, Switzerland

REFERENCES:
- [Derived] Atila C, Holze F, Murugesu R, Rommers N, Hutter N, Varghese N, Sailer CO, Eckert A, Heinrichs M, Liechti ME, Christ-Crain M. Oxytocin in response to MDMA provocation test in patients with arginine vasopressin deficiency (central diabetes insipidus): a single-centre, case-control study with nested, randomised, double-blind, placebo-controlled crossover trial. Lancet Diabetes Endocrinol. 2023 Jul;11(7):454-464. doi: 10.1016/S2213-8587(23)00120-1. Epub 2023 May 13. PMID 37192642